CLINICAL TRIAL: NCT05456607
Title: Optimizing Digital Behavioral Treatment for Co-occurring Insomnia and Depression
Brief Title: Digital CBT for Insomnia and Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of South Florida (Other); Harvard University (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Wilfred Pigeon, PhD, Professor of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00007379
Record Dates: First submitted 2022-07-05; First posted 2022-07-13 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Depression; Insomnia
Keywords: cognitive behavioral therapy; digital intervention; depression; insomnia
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (Active Comparator): Online Mood Monitoring for 12 weeks
  Interventions: Behavioral: Mood Monitoring
- Single Insomnia Treatment (Experimental): Cognitive-behavioral therapy for insomnia delivered in a self-managed online format (computer or phone app) with access to a coach. Duration of access for 12 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Single Depression Treatment (Experimental): Cognitive-behavioral therapy for depression delivered in a self-managed online format (computer or phone app) with access to a coach. Duration of access for 12 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Depression
- Sequenced Depression and Insomnia Treatment (Experimental): Cognitive-behavioral therapy for depression followed by cognitive-behavioral therapy for insomnia each delivered in a self-managed online format (computer or phone app) with access to a coach. Duration of access to the depression treatment only for 4 weeks after which the access to the insomnia treatment is also made available. Total duration of access for 12 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Behavioral: Cognitive Behavioral Therapy for Depression
- Sequenced Insomnia and Depression Treatment (Experimental): Cognitive-behavioral therapy for insomnia followed by cognitive-behavioral therapy for depression each delivered in a self-managed online format (computer or phone app) with access to a coach. Duration of access to the insomnia treatment only for 4 weeks after which the access to the depression treatment is also made available. Total duration of access for 12 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Behavioral: Cognitive Behavioral Therapy for Depression

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia consists of the standard features of this well-established insomnia treatment that will be delivered in this study via a mobile optimized web app. Participants also have access to an intervention coach/guide as needed.
  Other Names: CBT-I
  Arms: Sequenced Depression and Insomnia Treatment; Sequenced Insomnia and Depression Treatment; Single Insomnia Treatment
Behavioral: Cognitive Behavioral Therapy for Depression — Cognitive Behavioral Therapy for Depression consists of the standard features of this well-established depression treatment that will be delivered in this study via a mobile optimized web app. Participants also have access to an intervention coach/guide as needed.
  Other Names: CBT-D
  Arms: Sequenced Depression and Insomnia Treatment; Sequenced Insomnia and Depression Treatment; Single Depression Treatment
Behavioral: Mood Monitoring — The mood monitoring intervention is based on mood tracking principles in broader mood management interventions, but without any psychoeducational content or cognitive-behavioral exercises. Instead, participants will get access to a mobile optimized web app that allows users to enter their mood, tag related events, and view trends over time to raise awareness of how activities influence certain mood states.
  Arms: Control

SUMMARY:
This study has two primary objectives, each of which addresses critical clinical and research gaps for individuals who have co-occurring insomnia and depression. The first objective is to address whether sequential treatment of insomnia and depression is superior to a single treatment for either depression or for insomnia, and if so, which treatment sequence is optimal. The second objective is to determine if there are heterogeneity of treatment effects; that is, variation in which interventions are best for which individuals, and if so, to develop and individualized intervention rule to better match individuals with the treatment that is most likely to lead to the best outcomes. A large randomized trial will be conducted to meet these objectives.

DETAILED DESCRIPTION:
Although efficacious behavioral treatments like cognitive behavioral therapy for insomnia (CBT-I) and for depression (CBT-D) exist for insomnia and depression disorders, their impact on co-occurring symptoms can be modest and residual symptoms often remain. In addition, scalable versions of these interventions (like computer accessible or phone app versions) are needed for U.S. military Veterans who lack access to first-line interventions because of rural or other resource-limited environments. Finally, little is known about heterogeneity of treatment effects; that is, variation in which interventions are best for which individuals. This comparative effectiveness trial is designed to develop an an individualized intervention rule to match the right digital intervention to the right person with co-occurring insomnia and depression.

The study will use digital versions of CBT-I and CBT-D found to be efficacious for their intended target. A total of 1,500 participants who are Veterans with both insomnia and depression will be randomized with equal allocation to five study arms: two single interventions (CBT-I or CBT-D); two sequenced interventions (CBT-I+D or CBT-D+I); and a mood monitoring condition that will serve as the control group. Assessments occur at baseline, mid-treatment, post-treatment, at 3-month and 6-month follow-ups. The primary endpoint will be remission of both depression and insomnia at 3 months following the 12 week intervention period. All study activity will be conducted remotely including recruitment, treatment delivery and assessments, so that participants can be recruited nationwide.

The study will estimate average treatment effects on insomnia and depression remission at 3-months post-treatment (primary outcome) and 6-month maintenance of remission as well as treatment response. Significantly higher remission and response rates for sequenced rather than single interventions and lowest for the mood monitoring control condition are expected. Because variation in which interventions are best for which individuals are expected, study investigators will develop and evaluate an individualized intervention rule to determine an optimal approach for each participant in promoting 3-month remission of both disorders. A cutting-edge ensemble machine learning method will be used to do this. In a companion, subsequent trial with a new cohort of 800 participants, the investigators will evaluate whether assigning participants to a treatment condition via the individualized intervention rule is superior to simple randomization that does not consider individual factors in the treatment decision. This subsequent trial will be registered as a separate clinical trial, but will refer back to this current trial.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* U.S. Military Veterans
* endorse depression (Patient Health Questionnaire-depression score > 10)
* endorse insomnia (Insomnia Severity Index score > 10).

Exclusion Criteria are limited in accordance with real world effectiveness trials, but will include:

* pregnancy
* history of bipolar disorder
* history of psychosis
* current use of anti-psychotic medications or mood stabilizers (e.g., lithium)
* current suicidal ideation with active intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Dual Remission of Depression and Insomnia | 3 Months post-treatment
  The proportion of participants achieving dual remission in each study arm with Depression Remission defined as a total score of < 5 on the Patient Health Questionnaire (PHQ-9) and Insomnia Remission defined as a total score of < 8 on the Insomnia Severity Index (ISI).

SECONDARY OUTCOMES:
Depression Response | 3 Months post treatment
  The proportion of participants achieving a Depression treatment response defined as a ≥ 5 point reduction in the total PHQ-9 score
Insomnia Response | 3 Months post treatment
  The proportion of participants achieving an Insomnia treatment response defined as a ≥ 8 point reduction in the total ISI score

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred Pigeon, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Sleep Research Laboratory, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be submitted to a data repository: the Inter-university Consortium for Political and Social Research (ICPSR) data repository at the University of Michigan for secondary analysis.
Supporting Information: Study Protocol
Time Frame: A final dataset and codebook will be submitted to the the Inter-university Consortium for Political and Social Research (ICPSR) at the conclusion of the study and will remain available in accordance with ICPSR guidelines.
Access Criteria: Access criteria will be in accordance with the policies set forth by the data repository, the Inter-university Consortium for Political and Social Research (ICPSR), which are available at: https://www.icpsr.umich.edu/web/pages/datamanagement/lifecycle/access.html

REFERENCES:
- [Derived] Pigeon WR, Bishop TM, Bossarte RM, Schueller SM, Kessler RC. A two-phase, prescriptive comparative effectiveness study to optimize the treatment of co-occurring insomnia and depression with digital interventions. Contemp Clin Trials. 2023 Sep;132:107306. doi: 10.1016/j.cct.2023.107306. Epub 2023 Jul 28. PMID 37516163